CLINICAL TRIAL: NCT03257982
Title: A Feasibility Study of Patient Self-Managed Brain-computer Interface Functional Electrical Stimulation (BCI-FES) Hand Therapy for Spinal Cord Injured Patients
Brief Title: Patient Self-managed BCI-FES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Glasgow (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: GN17NE402
Record Dates: First submitted 2017-08-16; First posted 2017-08-22 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Spinal Cord Injuries
Keywords: Brain-computer interface; Functional electrical stimulation
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BCI-FES hand therapy (Experimental): BCI-FES hand therapy sessions (set up and use of system)
  Interventions: Procedure: BCI-FES hand therapy

INTERVENTIONS:
Procedure: BCI-FES hand therapy — BCI-FES rehabilitation therapy of the upper limb

SUMMARY:
This study aims to assess the feasibility of therapist-caregiver-patient training to use BCI and FES technology with a view to the inexpensive equipment eventually being used for home use by tetraplegic patients as a continuing rehabilitation method for sub-acute patients discharged from hospital.

DETAILED DESCRIPTION:
Spinal Cord Injury (SCI) affects a person's ability to move and feel sensation in the body. People with injury around the neck, suffer from tetraplegia, which affects function of both upper and lower limbs. Although these patients often have a caregiver, their main priority is to regain some upper limb function to increase independence. About half of patients with tetraplegia have an incomplete injury, i.e. have some sensation and control of muscles preserved. Natural recovery takes about a year and is typically accompanied by intense physical therapy while patients are in a hospital. Patients spend on average 4 months in hospital and, once they go home, there are very limited options for further therapy, in particular those living in rural areas.

This study will test the feasibility of patient and caregiver self-managed hand therapy based on the combination of brain computer interface (BCI) and functional electrical stimulation (FES). BCI is a system which consists of an electroencephalographic device (EEG), a computer and software that can analyse EEG while it is being recorded. To ensure that the knowledge stays within hospital, occupational therapists will first be trained who will then train patients and caregivers. The BCI-FES therapy is based on a previous clinical study with hospitalised patients, in which a researcher administered the therapy. In this study, a portable BCI-FES system will be used with an inexpensive consumer BCI, which is designed for non-professionals. The primary objective is to assess whether it is feasible for caregivers and patients to learn to operate the portable BCI-FES system on their own within 5 training sessions. The secondary objectives are to collect feedback from patients and therapists of their views via semi-structured interviews and questionnaires; to assess how stable the system parameters (EEG parameters, electrode location, FES stimulation parameters)are over time; to assess whether there is any functional and neurological recovery.

ELIGIBILITY:
Inclusion Criteria:

Patients

* being within a year post-injury
* has a caregiver willing to commit their time to the study
* normal or corrected to normal vision
* no history of brain disease or injury
* incomplete injury at level C2 to C7
* minimum computer literacy
* understands spoken and written English

Occupational therapists

* already has experience in providing occupational therapy to spinal cord injured people
* familiar with using FES on patients

Caregivers

* able and willing to commit time to the study
* minimum computer literacy
* possess mobile phone with a camera or are allowed to use patient's mobile phone with a camera for taking photos of the experimental setup (to remind themselves)
* understands spoken and written English

Exclusion Criteria:

Patients

* presence of neurological problem which may distort brain signal recording (e.g. epilepsy, Parkinson's disease, multiple sclerosis)
* presence of cognitive impairments which would prevent patients or caregivers from understanding the task
* inability to sit for 2 hours
* general poor health due to secondary consequences of injury
* any condition that would be contraindicative of using FES (pacemakers, sensitive skin/sores over areas where electrodes should be applied, pregnancy)

Occupational therapists

* unable to commit sufficient time to the study
* cannot learn to setup BCI-FES within 30 min within 4 hourly training sessions

Caregivers

* cannot be present for all five therapy sessions

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-01-25 (Actual); Primary Completion 2019-03-14 (Actual); Study Completion 2019-03-14 (Actual)

PRIMARY OUTCOMES:
Successful training for operation of BCI-FES system | 2 months
  Number of times patients/caregivers successfully operate BCI-FES system within 30 min

SECONDARY OUTCOMES:
System reliability | 2 months
  Number of times patients manage to activate the BCI-FES system
Time taken to use system | 2 months
  Average time required to accomplish BCI-FES therapy (excluding setup time)
NASA task load index | 2 months
  Score from National Aeronautics and Space Administration (NASA) Task Load Index questionnaire
Psychological Effect of Assistive Devices | 2 months
  Score of Psychological Effect of Assistive Devices questionnaire
Quebec User Evaluation of Satisfaction with Assistive Technology | 2 months
  Score of Quebec User Evaluation of Satisfaction with Assistive Technology questionnaire
Grip strength | Baseline and 2 months
  Change in grip strength
Hand range of motion | Baseline and 2 months
  Change in hand range of motion

CONTACTS AND LOCATIONS:
Overall Officials: Aleksandra Vuckovic, BEng MSc PhD, Study Director — University of Glasgow
Locations (1):
- Queen Elizabeth National Spinal Injuries Unit, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zulauf-Czaja A, Al-Taleb MKH, Purcell M, Petric-Gray N, Cloughley J, Vuckovic A. On the way home: a BCI-FES hand therapy self-managed by sub-acute SCI participants and their caregivers: a usability study. J Neuroeng Rehabil. 2021 Feb 25;18(1):44. doi: 10.1186/s12984-021-00838-y. PMID 33632262